CLINICAL TRIAL: NCT00009542
Title: Evaluation of the Effect of Kava on Drug Metabolism Enzymes and EEG Measured Beta Amplitude
Brief Title: Effects of Kava on the Body's Elimination of Caffeine and Dextromethorphan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010059; 01-CC-0059
Record Dates: First submitted 2001-01-27; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-01

CONDITIONS: Healthy
Keywords: Caffeine; Cytochrome P 450; Dextromethorphan; Herbal; Interactions; Alternative Therapy; Healthy Volunteer; Kava

INTERVENTIONS:
Drug: kava (Piper methysticum)

SUMMARY:
This study will examine how kava-a widely used herbal remedy-may affect the body's elimination of other medicines. Many people take kava to reduce anxiety or cause sedation. Since this product is considered a food supplement and not a drug, it is not subject to the rigorous pre-market testing required for prescription and over-the-counter (OTC) drugs. As a result, information has not been collected on possible interactions between kava and other medications. This study will look at how kava affects the elimination of caffeine-a compound commonly found in chocolate, coffee, tea and soft drinks-and dextromethorphan-an OTC cough suppressant.

Normal healthy volunteers 21 years of age or older may be eligible for this 30-day study. Candidates will provide a medical history and undergo a physical examination and routine blood tests. Women of childbearing age will have a urine pregnancy test.

Study participants will not drink alcoholic beverages or take any medications (except those given in the study) for 2 weeks prior to the study and throughout its duration. In addition, they will abstain from caffeine, grapefruit and grapefruit juice and charbroiled foods for at least 72 hours before and throughout each study day that urine is collected.

On day 1 of the study, study subjects will take one dose each of caffeine and dextromethorphan at 4:00 P.M.. They will empty their bladder before the dosing and then collect all their urine after the dosing for the rest of the day and including the next mornings first urine. They will bring the urine samples to the Clinical Center when the collection is complete. This procedure will be repeated 1 week later (study day 8). After the second urine collection is completed, subjects will take 200 milligrams of kava 3 times a day for 21 days. On study day 29 (after 21 days of kava), subjects will repeat the dextromethorphan and caffeine dosing and urine collection described above, while continuing to take kava.

Subjects will have an electroencephalograph (EEG) done before starting kava and again at the end of kava (study day 30). For this procedure, several electrodes (metal cups attached to wires) are secured to the scalp with a glue-like substance. A conductive gel fills the space between the electrode and the scalp to ensure good contact. The electrodes will remain in place for about 2 hours and then removed. The subject lies quietly on a bed during the EEG recording.

Participation in the study will end with another physical examination and blood tests following the second EEG and urine collection.

DETAILED DESCRIPTION:
Kava (piper methysticum) is a complementary or alternative medication used for purported anxiolytic and sedative effects. Despite its widespread use there is no data regarding potential for drug interactions or its effects on the electroencephalogram. The purpose of this study is to determine the effect of administration of kava for 3 weeks on the activity of cytochrome p450, 1A2, 2D6, 3A4; NAT2, and XO. Additionally, the effect of kava on EEG measured beta amplitude will be evaluated. Fifteen healthy volunteers will undergo enzyme activity phenotyping by ingesting 2 mg/kg of caffeine and 30 mg of dextromethorphan followed by an overnight urine collection. Following completion of two separate baseline evaluations, separated by 1 week, subjects will then take 1 capsule containing 60 mg of kavalactones three times daily for 3 weeks. Following 3 weeks of therapy subjects will undergo repeat enzyme activity phenotyping as described previously. Enzyme activity following 3 weeks of kava will be compared to pre-treatment values to characterize the magnitude of inhibition and/or induction of CYP1A2, CYP2D6, CYP3A4, NAT2, and XO activity. Additionally, subjects will have EEG testing performed to evaluate the effect of kava on beta amplitude. EEG's will be performed the day before the first baseline phenotyping procedure and then following three weeks of kava (the day before the final phenotyping procedure). Beta amplitude following three weeks of kava will be compared to pre-treatment values to evaluate the magnitude of pharmacodynamic effect. The results of this study will be used to facilitate the development of protocols to evaluate the magnitude of interactions between clinically relevant traditional medications and kava as well as studies to compare the pharmacologic effect of kava to the effects of benzodiazepines.

ELIGIBILITY:
Male or female

Healthy by medical history and physical exam

Age greater than 21 years old

No concurrent medications

Non-smoker (for at least 6 months if prior history of smoking)

Laboratory values within the following guidelines:

AST/SGOT less than or equal 1.5 X ULN

Bilirubin less than or equal 1.5 X ULN

Serum creatinine less than or equal ULN

Hemoglobin less than 10 g/dl

Females of child bearing potential must be using a reliable form of birth control other than hormonal contraceptives

Ability to abstain from caffeine containing foods/beverages, ethanol, grapefruit or grapefruit juice and charbroiled foods for 72 hours prior to, and the day of, phenotyping procedures.

Normal EEG during baseline testing.

No patients using concomitant therapy with other inhibitors or inducers of cytochrome P-450 mediated drug metabolism within 30 days of study.

No patients with inability to remain free of chronic medications and alcohol for atleast 2 weeks prior to and during the study.

Presence of renal, hepatic, cardiovascular, hematologic, neurologic, psychiatric, or respiratory disease or any other condition that may interfere with the interpretation of the study results or not be in the best interests of the subject in the opinion of the investigator.

Positive urine pregnancy test.

The presence of persistent diarrhea or malabsorption that would interfere with the patient's ability to adequately absorb drug.

Drug or alcohol use that may impair safety or adherence.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2001-01; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Elion RA, Cohen C. Complementary medicine and HIV infection. Prim Care. 1997 Dec;24(4):905-19. doi: 10.1016/s0095-4543(05)70316-x. PMID 9386262
- [Background] Israel D, Youngkin EQ. Herbal therapies for perimenopausal and menopausal complaints. Pharmacotherapy. 1997 Sep-Oct;17(5):970-84. PMID 9324185
- [Background] Eisenberg DM, Davis RB, Ettner SL, Appel S, Wilkey S, Van Rompay M, Kessler RC. Trends in alternative medicine use in the United States, 1990-1997: results of a follow-up national survey. JAMA. 1998 Nov 11;280(18):1569-75. doi: 10.1001/jama.280.18.1569. PMID 9820257